CLINICAL TRIAL: NCT02245282
Title: Contrast Enhanced MRI of the Prostate
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Garzotto, MD, Professor, OHSU Knight Cancer Institute
Other Study IDs: IRB00010345; 1R44CA180425 (NIH)
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prostate cancer detection and disease progression monitoring relies on systematic multi-core biopsies. Minimal invasive imaging capacities for lesion targeting and monitoring are badly needed. The purpose of this study is to determine if a new MRI technique can identify and monitor prostate disease progression. If so biopsy core number can be reduced to as small as one, and frequency for biopsy repeat can be reduced. The new technique is about a new way of analyzing the pictures taken as part of prostate MRI exam. This part is called dynamic contrast-enhanced MRI. It involves an injection of contrast reagent (or dye) through the arm vein during a time period when prostate MRI pictures are continuously taken.

DETAILED DESCRIPTION:
The aim of the study is to perform contrast-enhanced (CE) magnetic resonance imaging (MRI) at OHSU on subjects with diagnosed prostate cancer. This pilot project will study 20 subjects prior to their next scheduled clinical procedures (biopsy or radical prostatectomy). Data from this project will be used to explore new capabilities of the software platform developed under current SBIR funding. CE-MRI will involve the use of an extracellular (Gadolinium based, Gd) contrast agent. When Gd is used, (dynamic-contrast-enhanced) DCE-MRI signal intensity time-course data will be analyzed analytically using the so called "shutter-speed" paradigm which takes into account of the effects of finite water exchange kinetics. Region of interest (ROI) and high resolution (~millimeter) parametric maps of pathophysiologic quantities, such as tumor vessel permeability, tumor perfusion, extracellular extravascular volume fraction, will be generated from the DCE-MRI data. All parameters will be compared to literature results for software validation and correlated with pathology for clinical potential.

ELIGIBILITY:
Inclusion Criteria:

* Men, age >18 years.
* Any patient scheduled for prostate biopsy repeat or radical prostatectomy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who would be normally excluded from undergoing an MRI examination - patients with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field.
* Patients who are unable to cooperate for an MRI exam.
* Major surgery within a month of enrollment.
* Prostate biopsy six weeks prior to enrollment.
* Subject-reported reaction to gadolinium contrast reagent.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 subjects will be studied under this protocol. Subjects will be selected from patients scheduled for prostate biopsies with known prostate lesions. Subjects will also be recruited from prostate cancer patients who choose radical prostatectomy as disease management plan. The research project will be introduced to a potential subject by a urologist at OHSU. If interested, the subject will then be contacted through phone to participate in the study by an investigator or a research assistant on the research team.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Prostate Cancer Detection and Aggressiveness Monitoring by Contrast Enhanced MRI | within 60 days after MRI data collection

CONTACTS AND LOCATIONS:
Overall Officials: Mark Garzotto, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Advanced Imaging Research Center, OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared to Imbio LLC